CLINICAL TRIAL: NCT00272467
Title: A Comparative Study on the Healing Effects of Rebamipide and Omeprazole in Helicobacter Pylori-positive Gastric Ulcer After Eradication Therapy
Brief Title: Healing Effects of Rebamipide and Omeprazole in Helicobacter Pylori-positive Gastric Ulcer After Eradication Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka International Asia Arab (Industry)
Collaborators: Zhejiang Otsuka Pharmaceutical Co., Ltd. (Industry); Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OIAAMCTIVK205
Record Dates: First submitted 2006-01-04; First posted 2006-01-06 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Stomach Ulcer
Keywords: Helicobacter pylori; Stomach ulcer; Rebamipide; Omeprazole
MeSH Terms: conditions — Stomach Ulcer | interventions — rebamipide; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rebamipide (Experimental): 1. Dosage (1) The eradication therapy period (for all cases) Amoxicillin 2,000mg/day, clarithromycin 1,000 mg/day and omeprazole 40 mg/day. b.i.d. (morning and evening), oral administration. (2) The ulcer treatment period (on a double-blind basis) Rebamipide 100mg, t.i.d. (before breakfast, evening, before bed).
  2. Drug period (1) The eradication therapy period: 1 week (2) The ulcer treatment period: 7 weeks
  Interventions: Drug: Rebamipide
- Omeprazole (Active Comparator): 1. Dosage (1) The eradication therapy period (for all cases) Amoxicillin 2,000mg/day, clarithromycin 1,000 mg/day and omeprazole 40 mg/day. b.i.d. (morning and evening), oral administration. (2) The ulcer treatment period (on a double-blind basis) omeprazole 20mg, once daily (before breakfast)
  2. Drug period (1) The eradication therapy period: 1 week (2) The ulcer treatment period: 7 weeks
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Rebamipide — 1. Brand name: Mucosta® Tab.
  2. Generic name: Rebamipide.
  3. Chemical name:
     (±)-2-(4-chlorobenzoylamino)-3-[2(1H)-quinolinon-4-yl]propionic acid.
  4. Formulation: Tablet (White, film-coated tablet).
  5. Strength: One tablet contains rebamipide 100mg.
  6. Storage condition: 15℃~25℃.
  7. Manufacturer: Korea Otsuka Pharmaceuticals
  Other Names: Mucosta
  Arms: Rebamipide
Drug: Omeprazole — 1. Brand name: Losec® Cap.
  2. Generic name: Omeprazole.
  3. Chemical name:
  5-melthoxy-2-{{{4-melthoxy-3.5-dlmethyl2-pyridinyl}methyl}sulp- hinyl}-1H-benzimidazole sodium. 4) Formulation: Capsule. 5) Strength: One capsule contains omeprazole 20mg. 6) Storage condition: 15℃~25℃. 7) Manufacturer: AstraZenaca Korea.
  Other Names: Losec
  Arms: Omeprazole

SUMMARY:
The purpose of this study is to evaluate the ulcer healing efficacy of rebamipide in comparison with omeprazole in Helicobacter pylori-positive gastric ulcer after eradication therapy.

DETAILED DESCRIPTION:
This study is designed to evaluate the ulcer healing efficacy of rebamipide administered following the eradication therapy in comparison with the well known PPI, omeprazole. This is a double-blind, comparative study which is expected to prove the role of rebamipide in gastric ulcer healing after the eradication therapy. This study may contribute to further clinical research on a new type of ulcer treatment by looking at the treatment modality based on the enhancement of defensive factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 or older at the time of writing the informed consent
* H. pylori-positive patient.
* Patients who are diagnosed with gastric ulcer by endoscopy and have the following ulcer characteristics; Non-scarring ulcer (stage A1, A2, H1, H2 according to the Sakita-Miwa classification), Single ulcer, Ulcer size of 5 to 20mm in diameter

Exclusion Criteria:

* Patients who previously underwent H. pylori eradication therapy
* Malignant gastric ulcer
* Linear ulcer
* Patients with history of upper GI tract resection or vagotomy
* Patients with continuous NSAIDs use within 4 weeks prior to study initiation
* Patients with ulcer complications including perforation or pyloric stenosis
* Gastric ulcer prone to bleeding (e.g. exposed blood vessels at ulcer base)
* Patients with infectious mononucleosis
* Patients with known hypersensitivity to penicillin, clarithromycin, omeprazole, amoxicillin or rebamipide
* Patients on medications such as terfenadine or pimozide which are contraindicated with clarithromycin usage
* Pregnant or possibly pregnant women, lactating women, or those with a plan to conceive during this study
* Blood test results of Hb ≤ 8.0 g/dl, platelet ≤50,000 /㎕, total WBC ≤ 4000/㎕ or ≥ 10,000/㎕, and with serum test results showing the levels of AST, ALT, ALP, LDH, BUN, and creatinine exceeding twice the normal range of respective institution.
* Other patients deemed not eligible for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2005-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Gastric ulcer healing rate | at 12 weeks after the initial administration of the study medication
  Rebamipide showed 81.5~87.8% of gastric ulcer healing rate which was not inferior to 82.5~87.8% healing rate of Omeprazole.

SECONDARY OUTCOMES:
Gastric ulcer healing rate in cases with successful H.pylori eradication and H.pylori eradication failure (12 weeks after administration of the study medication.) | at 12 weeks after the initial administration of the study medication
Serum gastrin level | at 8 and 12 weeks after the initial administration of study medication
Economical efficiency | drug cost/effect ratio
  Rebamipide was more cost effective than Omeparzole for 7 weeks of gastric ulcer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ho Kim, M.D., Principal Investigator — Asan Medical Center, Ulsan University
Locations (7):
- China (5):
  - The 1st Affiliated hospital - Zhongshan Univ., Guangzhou, Guangdong
  - Nanfang Hospital - Nanfang Medical Univ., Guangzhou, Guangdong
  - Xijing Hospital - The 4th Military Medical Univ, Xi’an, Shanxi
  - The 1st Affiliated Hospital - Medical School of Zhejiang Univ., Hangzhou, Zhejiang
  - Ren-Ji Hospital - Shanghai Second Medical Univ., Shanghai
- South Korea (2):
  - Korea University Ansan Hospital, Ansan
  - Severance Hospital, Seoul National University, Seoul